CLINICAL TRIAL: NCT02530593
Title: QoLiCOL - Quality of Life in Colon Cancer
Acronym: QoLiCOL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Principal Investigator, Sahlgrenska University Hospital
Other Study IDs: QoLiCOL
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Colonic Neoplasm
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with colon cancer: All patients presenting with a newly diagnosed colon cancer regardless of tumour stage
  Interventions: Behavioral: There is no intervention, only observation

INTERVENTIONS:
Behavioral: There is no intervention, only observation

SUMMARY:
All patients presenting at participating hospitals during the recruitment period with a newly diagnosed colon cancer, regardless of stage and planned treatment, will be eligible for inclusion. They will answer a questionnaire on health related quality of life, physical symptoms, functional impairments and socioeconomic status at diagnosis and after 12, 36 months. Clinical data including recurrence, survival, surgical treatment, oncologic result (pathology report) and adjuvant treatment will be collected from the Swedish ColoRectal Cancer Registry (SCRCR)

DETAILED DESCRIPTION:
QoLiCOL is an explorative, prospective, longitudinal, non-interventional, international, multicenter study of health-related quality of life, physical symptoms, functional impairments and socioeconomic burden in colon cancer patients. All patients presenting at participating hospitals during the recruitment period with a newly diagnosed rectal cancer, regardless of stage and planned treatment, will be eligible for inclusion. Patients will be followed for 3 years. They will be asked to answer questionnaires at three different time points during follow-up: at diagnosis and after 12 and 36 months. Clinical data, including recurrence, surgical treatment, oncologic result (pathology report) and adjuvant treatment will be collected from the national quality registry for rectal cancer in Denmark and Sweden. As these registries differ in some areas between the countries, additional data will be collected through short CRF:s.

ELIGIBILITY:
Inclusion Criteria:

* Colon cancer newly diagnosed.
* Planned treatment presented

Exclusion Criteria:

* No Colon cancer diagnosis,
* below 18 years of age,
* no informed consent or withdrawn informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer prior to treatment initiation.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-06; Primary Completion 2022-11 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
QoL in colon cancer patients | 3 years
  The primary end-point is to describe QoL, symptoms and functional impairments in an unselected population of colon cancer patients

SECONDARY OUTCOMES:
Generate basic descriptive data of the patient population, such as demography, socioeconomic data, disease stage at diagnosis, type of treatment, recurrence and survival | 3 years
Compare differences in QoL between patients with different tumour levels | 3 years
Detect differences in QoL in patients over time after colon cancer treatment | 3 years
Evaluate the effect of complications after colon cancer surgery on the patients socioeconomic situation | 3 years
Evaluate the effect of coping strategies on QoL after initiated treatment | 3 years
Describe patient expectations at diagnosis of colon cancer | 3 years
Identify differences in QoL between patients in different groups regarding gender, age and education level | 3 years
Analyse how clinical factors like oncologic result of operation, morbidity, recurrence and survival influence QoL | 3 years
Identify areas of improvement in treatment and patient care | 3 years
Enable initiation interventional studies when appropriate | 3 years
Analyse health economy aspects of QoL and morbidity in the patient population | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — SSORG
Locations (1):
- Sahlgrenska University Hospital/Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sandberg SJ, Park JM, Tasselius VA, Angenete E. Bowel Dysfunction After Colon Cancer Surgery: A Prospective, Longitudinal, Multicenter Study. Dis Colon Rectum. 2024 Oct 1;67(10):1322-1331. doi: 10.1097/DCR.0000000000003358. Epub 2024 Jun 20. PMID 38902840
- [Derived] Ehrencrona C, Li Y, Angenete E, Haglind E, Franzen S, Grimby-Ekman A, Bock D. Do beta-blockers reduce negative intrusive thoughts and anxiety in cancer survivors? - An emulated trial. BMC Cancer. 2024 Apr 11;24(1):447. doi: 10.1186/s12885-024-12236-3. PMID 38605350